CLINICAL TRIAL: NCT05232890
Title: Hydroponic Cultivation: a New Dietary Frontier in Systemic Nickel Allergy Syndrome - a Double Blind, Randomized, Controlled, Cross-over, Clinical Trial on the Use of Hydroponic Cultivated Tomato Sauce
Brief Title: Hydroponic Cultivation in Systemic Nickel Allergy Syndrome
Acronym: DATTERINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Eleonora Nucera, Head of Allergy Unit, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ID3643
Record Dates: First submitted 2021-11-17; First posted 2022-02-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Food Allergy; Food Hypersensitivity; Nickel Sensitivity
Keywords: Systemic Nickel Allergy Syndrome; Hydroponic cultivation; Tomato; Quality of life; Intestinal permeability
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: At enrollment, patients are randomized to one of the following study groups: Group A and Group B:
  * Treatment arm A: daily intake of minimum 100ml - maximum 200ml of 100% Italian datterino tomato puree deriving from hydroponic technology (soilless), contained in a 720ml bottle.
  * Treatment arm B: daily intake of minimum 100ml - maximum 200ml of 100% Italian datterino tomato puree deriving from conventional cultivation, contained in a 720ml bottle.
  After this initial treatment phase, both study groups follow a 2-week wash-out period, following a low-nickel diet.
  At the end of the wash-out phase, the two groups cross-over. Therefore, Group A is assigned to treatment arm B, and vice versa, for a period of 12 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study product and the comparator product are provided in identical packaging, the labeling shows the randomization number which, however, only the Outcomes Assessor is able to refer to the type of treatment assigned. The organoleptic characteristics of the two products are as similar as possible. The instructions given to patients regarding the preparation and consumption of the products are the same for both products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Datterino tomato purée from hydroponic technology (Experimental): 100% Italian datterino tomato purée deriving from hydroponic technology (soilless) with particular characteristics such as nickel free and zero residue.
  Interventions: Other: Datterino tomato purée from hydroponic technology
- Datterino tomato purée from conventional cultivation (Active Comparator): 100% Italian datterino tomato purée deriving from conventional cultivation.
  Interventions: Other: Datterino tomato puree from conventional cultivation

INTERVENTIONS:
Other: Datterino tomato purée from hydroponic technology — Daily intake of minimum 100ml - maximum 200ml of 100% Italian datterino tomato puree deriving from hydroponic technology (soilless), contained in a 720ml bottle.
  Arms: Datterino tomato purée from hydroponic technology
Other: Datterino tomato puree from conventional cultivation — Daily intake of at least 100ml - maximum 200ml of 100% Italian datterino tomato puree deriving from conventional cultivation, contained in a 720 ml bottle.
  Arms: Datterino tomato purée from conventional cultivation

SUMMARY:
Oral intake of nickel (Ni) is capable of causing the onset of systemic disorders in patients with Systemic Allergy to Nickel Syndrome (SNAS), an emerging allergic condition. Given its ubiquitous age, it is not possible to completely eliminate Ni and, therefore, it is necessary to plan a low-content diet. However, due to various factors (such as variability of Ni concentration in the soil, individual foods, variability of dietary habits and daily menus, different intake of Ni contained in the water, different intake of kitchen utensils, simultaneous intake of other substances), a restrictive diet is difficult and socially discriminating with a strongly negative impact on the quality of life of these patients.

Hydroponic agriculture in a completely controlled, aseptic, artificial, soilless environment could be an alternative for patients suffering from SNAS with known and lower concentrations of metals than those deriving from conventional agricultural techniques, which are affected by the soil of origin and practices cultivation.

The primary outcome of the study is to evaluate the possible effects of taking tomato puree deriving from hydroponic agriculture compared to tomato puree from conventional cultivation in the subjective control of SNAS symptoms, in patients following a low-diet diet.

This is an interventional, randomized, double-blind, single-center crossover study involving a cohort of SNAS patients following a low-nickel diet for at least 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented diagnosis of SNAS: a) history of SNAS (coexistence of typical skin symptoms and gastrointestinal symptoms); b) positive nickel sulphate patch test; c) clinical improvement of at least 70% after 4-6 weeks of low-nickel diet; d) positivity of the oral challenge test with nickel sulphate.
* Age between 18 and 65 years.
* Written informed consent to participate in the study.
* Patients who are able to participate in all study procedures and to accept and comply with all study needs throughout the study, including the availability of suitable transportation and the time required to undergo all procedures. planned visits.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Patients diagnosed with organic diseases capable of affecting gastrointestinal symptoms (eg celiac disease, poorly controlled diabetes, scleroderma, chronic inflammatory bowel diseases). Lactose intolerance is not an exclusion criterion if the diagnosis has been made for more than 6 months and if the patient does not report adequate symptom relief after at least 6 months of a lactose-free diet.
* Patients who have been taking systemic probiotics, antibiotics or systemic corticosteroids within the past 30 days.
* Patients who have been taking antidepressant or anxiolytic drugs for less than a month. On the other hand, patients can be enrolled who have been taking the aforementioned drugs at a stable dosage for at least one month.
* Patients who abuse coffee, tea, coca cola and with a smoking habit.
* Patients with pacemakers because they cannot be subjected to bioimpedance analysis for the assessment of body composition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change of gastrointestinal symptoms control | Immediately after the intervention
  Average values of the scores relating to the individual SNAS symptoms as reported in the visual analogue scale (VAS) - Systemic Nickel Allergy Syndrome (SNAS) scale before and after taking each type of tomato sauce (hydroponic vs conventional).
  This scale includes values from a minimum of zero to a maximum of ten. Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Change of impact on quality of life - SF-36 | Change from baseline index at 12 and 26 weeks.
  Difference in mean scores on quality of life questionnaire Short Form 36 Items Health Survey (SF-36) before and after each planned dietary treatment (hydroponic vs conventional tomato).
  Each patient answers SF-36v2 (Italian version) questionnaire. It comprises 36-items measuring 8 dimensions of general QoL. Each question's score is coded, summed up, and transformed to a scale of 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).
Change of impact on quality of life - PGWBI | Change from baseline index at 12 and 26 weeks.
  Difference in mean scores on quality of life questionnaire Psychological General Well Being Index (PGWBI) before and after each planned dietary treatment (hydroponic vs conventional tomato).
  PGWBI consists of 22 questions, which deal with 6 factors (anxiety, depression, vitality, general health,self-control and well-being) constituting a global assessment. The response format is graded 1-6. This index includes values from a minimum of 0 to a maximum of 110. Higher scores indicate a better outcome.
Change of intestinal permeability | Change from baseline index at 12 and 26 weeks.
  Difference in mean values of serum zonulin (a biomarker of intestinal permeability) before and after each planned dietary treatment (hydroponic vs conventional tomato puree).
Change of beta-carotene | Change from baseline index at 12 and 26 weeks.
  Difference in the average values of beta-carotene [microg/dl] before and after each planned dietary treatment (hydroponic vs conventional tomato puree).
Change of Vitamin D | Change from baseline index at 12 and 26 weeks.
  Difference in the average values of Vitamin D [ng/ml] before and after each planned dietary treatment (hydroponic vs conventional tomato puree).
Change of hemoglobin | Change from baseline index at 12 and 26 weeks.
  Difference in the average values of hemoglobin [g/dl] before and after each planned dietary treatment (hydroponic vs conventional tomato puree).
Change of ferritin | Change from baseline index at 12 and 26 weeks.
  Difference in the average values of ferritin [ng/ml] before and after each planned dietary treatment (hydroponic vs conventional tomato puree).
Change of adherence | After 12 weeks, after 26 weeks.
  Cross-comparison between the percentages of weekly intake [average number of days per week] of tomato puree (hydroponic tomato puree before and conventional after versus conventional tomato puree before and hydroponic after).

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Nucera, Prof., MD, Principal Investigator — Catholic University of Sacred Heart; Angela Rizzi, MD, PhD, Principal Investigator — Catholic University of Sacred Heart; Antonio Gasbarrini, Prof., MD, Study Director — Catholic University of Sacred Heart
Locations (1):
- UOSD Allergologia e Immunologia Clinica, Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No